CLINICAL TRIAL: NCT03665532
Title: Unified Intervention to Impact HIV Care Continuum
Brief Title: Youth Engagement Study: Intervention to Increase HIV Treatment Engagement and Adherence for Young People Living With HIV
Acronym: YES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Mercer University (Other)
Responsible Party: Principal Investigator, Seth Kalichman, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H16-130
Record Dates: First submitted 2017-05-27; First posted 2018-09-11 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive 2-way texting (Experimental): Biweekly text message communications with counselors for problem solving
  Interventions: Behavioral: Youth Engagement in Services
- Passive text reminders (Active Comparator): Automated weekly text message health care reminders
  Interventions: Behavioral: Youth Engagement in Services

INTERVENTIONS:
Behavioral: Youth Engagement in Services — Brief phone coaching to enhance engagement, retention, and sustain adherence to HIV and substance use services for younger people living with HIV.

SUMMARY:
This pragmatic adaptive clinical trial will test the effects of a Stigma-Motivational-Decision intervention designed to increase HIV treatment engagement, retention, and medication adherence for substance using adolescents and young adults (AYA) living with HIV who are not in clinical care. The intervention uses a uniquely unified counseling approach at multiple points along the HIV continuum of care. The trial will use multiple modes of outreach including social media, passive media, clinic records, and chain referrals to seek and identify HIV positive AYA who are HIV untreated, under-dosed, or unsuppressed (HIV-U3). Participants will receive phone-delivered Stigma-Motivational-Decision counseling intervention sessions to achieve engagement or re-engagement in HIV care, treatment adherence and control of their HIV infection. Once viral control is achieved, participants will receive a low-cost approach to sustaining long-term retention in care and medication adherence.

DETAILED DESCRIPTION:
This pragmatic adaptive clinical trial will test the effects of a Stigma-Motivational-Decision intervention designed to increase HIV treatment engagement, retention, and antiretroviral (Art) medication adherence for substance using adolescents and young adults (AYA) living with HIV who are not in clinical care. The intervention uses a uniquely unified counseling approach at multiple points along the HIV continuum of care. In a first step, the study will use multiple modes of outreach including social media, passive media, clinic records, and chain referrals to seek and identify HIV positive AYA who are HIV untreated, under-dosed, or unsuppressed (HIV-U3). Identified AYA will be enrolled in a run-in to the trial to objectively confirm the following criteria for trial entry. In Step 2, Individuals who meet entry criteria -specifically - substance using HIV-U3 AYA - will be enrolled in a mobile health (mHealth) intervention to address substance use, HIV stigmas, medical care-related concerns, structural barriers, and other challenges to engaging youth in HIV care. Counseling will be provided weekly by cellphone until the time participants are receiving ART, adequately dosed on ART, and HIV suppressed within a maximum of 12 sessions (up to 3-months). The study will therefore determine the number of theory-based mHealth intervention sessions needed (minimally effective dose) for optimal treatment outcomes and the associated costs. Once engaged and optimally treated, Step 3 will conduct a randomized trial to test the comparative effects and cost effectiveness of two interventions to sustain long-term retention in care and medication adherence: (a) interactive text messaging with opportunities for ongoing supportive problem solving vs. (b) passive text message reminders. HIV positive AYA are likely to drop out of care because of known challenges such as substance use, social barriers such as stigma, and concerns regarding treatment. The 3-step study will use a single theory-based approach to determine the number of phone-delivered Stigma-Motivational-Decision counseling intervention sessions necessary to achieve engagement or re-engagement in HIV care, and will test the effects of a low-cost approach to sustaining long-term retention in care and medication adherence. The study will determine the minimally effective amount of counseling needed to engage substance using HIV positive AYA in care. The study will also test the effects of the counseling and text messaging interventions on maintaining HIV care retention, medication adherence, and HIV viral suppression over 18-months. The study will perform economic evaluations to determine the cost-effectiveness of the engagement-retention-adherence intervention and the effects of low-burden retention/adherence interventions to maintain retention in care and avoid relapse to non-adherence for AYA living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 years and 35 years
* HIV positive
* At least one of the following:

  * Active substance using
  * HIV untreated
  * Under-dosed with ART
  * HIV viral unsuppressed

Exclusion Criteria:

* Not HIV positive
* Younger than 16
* Older than 35 years of age

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
HIV suppression | up to 15 months after the baseline.
  Blood plasma derived HIV RNA

SECONDARY OUTCOMES:
Medication Adherence | up to 15 months after the baseline.
  Antiretroviral medication adherence assessed by unannounced phone pill counts

CONTACTS AND LOCATIONS:
Overall Officials: Seth C Kalichman, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Southeast HIV/AIDS Research & Evaluation Project, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiginton JM, Eaton LA, Earnshaw VA, Watson RJ, Kalichman SC. Socio-cognitive facilitators of ART-adherence among predominantly black sexual and gender minoritized persons living with HIV in Atlanta, Georgia: a latent profile analysis. J Behav Med. 2024 Dec;47(6):1012-1027. doi: 10.1007/s10865-024-00510-5. Epub 2024 Aug 31. PMID 39214949
- [Derived] Kalichman SC, Kalichman MO, Eaton LA. Phone-Delivered Intervention to Improve HIV Care for Young People Living With HIV: Trial to Inform Implementation and Utility. J Acquir Immune Defic Syndr. 2023 Nov 1;94(3):227-234. doi: 10.1097/QAI.0000000000003279. Epub 2023 Oct 13. PMID 37643392
- [Derived] Brousseau NM, Kalichman SC, Watson RJ, Eaton LA. Amphetamine use and its associations with antiretroviral adherence and viral load among sexual minority men and transgender women living with HIV. AIDS Care. 2023 Oct;35(10):1472-1479. doi: 10.1080/09540121.2023.2206096. Epub 2023 May 3. PMID 37139536
- [Derived] Kalichman SC, Eaton LA, Kalichman MO. Believing That It Is Hazardous to Mix Alcohol With Medicines Predicts Intentional Nonadherence to Antiretrovirals. J Acquir Immune Defic Syndr. 2022 Jun 1;90(2):208-213. doi: 10.1097/QAI.0000000000002933. PMID 35125476